CLINICAL TRIAL: NCT06911983
Title: Comparative Efficacy of Metformin and Berberine Among TCF7L2 (rs7903146) TT vs. CC Genotype Carriers With Type 2 Diabetes: A Pilot Randomized Clinical Study
Brief Title: Comparative Efficacy of Metformin and Berberine Among TCF7L2 (rs7903146) TT vs. CC Genotype Carriers With Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW026
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitis
Keywords: genetics; polymorphysm; supplements; berberine
MeSH Terms: interventions — Metformin; Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin Group (Active Comparator): Initial dose: 500 mg twice daily
  * Titration: increased to 1,000 mg twice daily by Week 2 if tolerated
  * Maximal dose: 2,000 mg/day
  Interventions: Drug: Metformin
- Berberine Group (Experimental): * Dose: 500 mg three times daily (1,500 mg/day total)
  * Formulation: standardized berberine HCl tablets
  * Duration: 12 weeks
  Interventions: Dietary Supplement: Berberine

INTERVENTIONS:
Drug: Metformin — Metformin • Initial dose: 500 mg twice daily • Titration: increased to 1,000 mg twice daily by Week 2 if tolerated • Maximal dose: 2,000 mg/day
  Arms: Metformin Group
Dietary Supplement: Berberine — Berberine
  * Dose: 500 mg three times daily (1,500 mg/day total)
  * Formulation: standardized berberine HCl tablets
  * Duration: 12 weeks
  Arms: Berberine Group

SUMMARY:
This pilot 12-week randomized open-label study compares metformin and berberine in newly diagnosed type 2 diabetes patients stratified by the TCF7L2 (rs7903146) genotype (TT vs. CC). The primary goal is to assess changes in HbA1c between metformin and berberine treated groups within each genotype. Secondary outcomes include fasting and postprandial glucose, insulin levels, HOMA-IR, body weight/BMI, lipid profile and adverse events.

The central hypothesis is that berberine, through its additional effect on TCF7L2-linked pathways, will provide superior glycemic control in high-risk TT carriers compared to metformin, whereas both treatments will yield comparable results in CC carriers. By enrolling only TT and CC genotypes, this study aims to estimate effect sizes and feasibility, guiding a future, larger-scale trial on genotype-tailored diabetes therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30-65 years;
* Newly diagnosed T2DM ≤1 year;
* Baseline HbA1c: 7.0-9.0% (53-75 mmol/mol);
* No prior use of antihyperglycemic agents or ≤4 weeks of usage;
* Willing to sign informed consent and undergo TCF7L2 genotyping;
* TT or CC genotype (rs7903146)

Exclusion Criteria:

* Severe comorbidities (hepatic, renal, cardiac dysfunction);
* Pregnancy or lactation;
* Known allergy or intolerance to metformin or berberine;
* Participation in another clinical trial within the last 3 months;
* TC genotype (excluded).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 12 weeks
  Change in HbA1c from baseline to Week 12 in each genotype group (TT or CC), comparing: TT + Berberine vs. TT + Metformin
Change in HbA1c from baseline (CC + Berberine vs. CC + Metformin) | 12 weeks

SECONDARY OUTCOMES:
Fasting Plasma Glucose change (FPG) | 12 weeks
Postprandial Glucose (PPG) change | 12 weeks
Serum Insulin Levels | 12 weeks
HOMA-IR change | 12 weeks
Body Weight in kg change | 12 weeks
Total Cholesterol change | 12 weeks
Triglycerides change | 12 weeks
LDL-C change | 12 weeks
HDL-C change | 12 weeks
Number of any adverce events | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Center for New Medical Technologies, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No